CLINICAL TRIAL: NCT02758171
Title: Bioequivalence of a Fixed Dose Combination Tablet of Empagliflozin/Linagliptin Compared With the Free Combination of Empagliflozin Tablet and Linagliptin Tablet in Healthy Male and Female Subjects (an Open-label, Randomised, Single-dose, Crossover Study)
Brief Title: Bioequivalence of a Fixed Dose Combination Tablet of Empagliflozin/Linagliptin Compared With the Free Combination of Empagliflozin Tablet and Linagliptin Tablet in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1275.21; 2015-004234-98 (EudraCT Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-02 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Linagliptin

ARMS (2):
- Empagliflozin+Linagliptin FDC (Experimental): One tablet fix dose combination (FDC)
  Interventions: Drug: Empagliflozin; Drug: Linagliptin
- Empagliflozin+Linagliptin single tablets (Active Comparator)
  Interventions: Drug: Empagliflozin; Drug: Linagliptin

INTERVENTIONS:
Drug: Empagliflozin
Drug: Linagliptin

SUMMARY:
The primary objective of this trial is to investigate the bioequivalence of one fixed dose combination tablet of empagliflozin/linagliptin (Test, T) compared with the free combination of one empagliflozin tablet and one linagliptin tablet (Reference, R) administered as single dose under fasted conditions.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure [BP], Pulse Rate [PR]), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and local legislation
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:
* Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device
* Sexually abstinent
* A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
* Surgically sterilised (including hysterectomy)
* Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH (Follicle Stimulating Hormone) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure [BP], Pulse Rate [PR] or Electrocardiogram [ECG]) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- FDC/Empagliflozin+Linagliptin: The subjects were administered one FDC (Fixed-Dose Combination) film-coated tablet containing 10 mg Empagliflozin and 5 mg Linagliptin orally with 240 mL of water after an overnight fast of at least 10 hours (h), as a single dose in the fasted state on Day 1 of Test treatment (T) in period 1, followed by one film-coated tablet containing 10 mg Empagliflozin (reference product 1) in combination with 1 film-coated tablet containing 5 mg Linagliptin (reference product 2) administered orally with 240 mL of water after an overnight fast of at least 10 h, as single doses in the fasted state on Day 1 of Reference treatment (R) in period 2.
  A wash-out period of at least 35 days was set following the drug administration in each period.
- Empagliflozin+Linagliptin/FDC: The subjects were administered one film-coated tablet containing 10 mg Empagliflozin (reference product 1) in combination with 1 film-coated tablet containing 5 mg Linagliptin (reference product 2) orally with 240 mL of water after an overnight fast of at least 10 h, as single doses in the fasted state on Day 1 of Reference treatment (R) in period 1, followed by one FDC film-coated tablet containing 10 mg Empagliflozin and 5 mg Linagliptin administered orally with 240 mL of water after an overnight fast of at least 10 h, as a single dose in the fasted state on Day 1 of Test treatment (T) in period 2.
  A wash-out period of at least 35 days was set following the drug administration in each period.
Period: Treatment Period 1
Arm/Group | FDC/Empagliflozin+Linagliptin | Empagliflozin+Linagliptin/FDC
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Wash-out
Arm/Group | FDC/Empagliflozin+Linagliptin | Empagliflozin+Linagliptin/FDC
Started | 28 | 28
Completed | 26 | 28
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other reason | 1 | 0
Period: Treatment Period 2
Arm/Group | FDC/Empagliflozin+Linagliptin | Empagliflozin+Linagliptin/FDC
Started | 26 | 28
Completed | 26 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This subject set included all subjects from the Randomised Set (RS) [ included all randomised subjects, whether treated or not] who were documented to have received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | FDC/Empagliflozin+Linagliptin | Empagliflozin+Linagliptin/FDC | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (9.7) | 38.9 (10.2) | 39.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz (Area Under the Concentration-time Curve of Empagliflozin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point)
Description: This outcome measure presents area under the concentration-time curve of Empagliflozin in plasma over the time interval from 0 to the last quantifiable data point.
  Time frame description: The time -1:00 hour (h) was approximate; the procedure was to be performed and completed within 2h before drug administration. PKS including participants with available data for AUC0-tz (area under the concentration-time curve of Empagliflozin in plasma over the time interval from 0 to the last quantifiable data point).
Time Frame: 1:00 [hour (h): minute] before drug administration and 0:20h, 0:40h, 1:00h, 1:30h, 2:00h, 2:30h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 24:00h, 34:00h, 48:00h, and 72:00h after drug administration.
Population: PharmacoKinetic parameter analysis Set (PKS): This subject set included all subjects from the TS who provided at least 1 primary or secondary PK parameter that was judged as PK evaluable and not affected by protocol violations relevant to the evaluation of PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- FDC (10 mg Empagliflozin and 5 mg Linagliptin): The subjects were administered one FDC film-coated tablet containing 10 mg Empagliflozin and 5 mg Linagliptin orally with 240 mL of water after an overnight fast of at least 10 hours (h), as a single dose in the fasted state on Day 1 of Test treatment (T).
- Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets: The subjects were administered one film-coated tablet containing 10 mg Empagliflozin (reference product 1) in combination with 1 film-coated tablet containing 5 mg Linagliptin (reference product 2) orally with 240 mL of water after an overnight fast of at least 10 h, as single doses in the fasted state on Day 1 of Reference treatment (R).
Arm/Group | FDC (10 mg Empagliflozin and 5 mg Linagliptin) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets
Number analyzed (Participants) | 55 | 54
nmol*h/L | 2550 (18.0) | 2510 (19.9)
Statistical Analysis 1: Comparison: FDC (10 mg Empagliflozin and 5 mg Linagliptin) vs Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets; The statistical model used was an Analysis of Variance (ANOVA) model on the logarithmic scale. This model included effects accounting for the following sources of variation: Sequence, subjects within sequences, period, and treatment. The effect subjects within sequences was considered as random, whereas the other effects were considered as fixed; Test type: Non-Inferiority or Equivalence — Bioequivalence acceptable range of 80.00% to 125.00%; p < 0.0001, ANOVA; Adjusted geometric mean (gMean) ratio = 101.71, 90% CI 2-sided [99.818 to 103.644], Standard Deviation 5.8 — The ratio [%] calculated as T [FDC (10 mg Empagliflozin and 5 mg Linagliptin)]/R [Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets]. Standard deviation is actually intra-individual geometric coefficient of variation (gCV) [%]

2. Primary Outcome: AUC0-72 (Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 to 72 Hours)
Description: This outcome measure presents area under the concentration-time curve of Linagliptin in plasma over the time interval from 0 to 72 hours.
  Time frame description: The time -1:00h was approximate; the procedure was to be performed and completed within 2h before drug administration. PKS including participants with available data for AUC0-72 (area under the concentration-time curve of Linagliptin in plasma over the time interval from 0 to 72 hours).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC (10 mg Empagliflozin and 5 mg Linagliptin) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets
Number analyzed (Participants) | 55 | 54
nmol*h/L | 281 (22.5) | 283 (23.3)
Statistical Analysis 1: Comparison: FDC (10 mg Empagliflozin and 5 mg Linagliptin) vs Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Bioequivalence acceptable range of 80.00% to 125.00%; p < 0.0001, ANOVA; Adjusted geometric mean (gMean) ratio = 99.39, 90% CI 2-sided [95.290 to 103.672], Standard Deviation 13.1 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Cmax (Maximum Measured Concentration of Empagliflozin Analyte in Plasma)
Description: This outcome measure presents maximum measured concentration of Empagliflozin analyte in plasma.
  Time frame description: The time -1:00h was approximate; the procedure was to be performed and completed within 2h before drug administration. PKS including participants with available data for Cmax (maximum measured concentration of Empagliflozin analyte in plasma).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | FDC (10 mg Empagliflozin and 5 mg Linagliptin) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets
Number analyzed (Participants) | 55 | 54
nmol/L | 370 (23.9) | 365 (23.9)
Statistical Analysis 1: Comparison: FDC (10 mg Empagliflozin and 5 mg Linagliptin) vs Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Bioequivalence acceptable range of 80.00% to 125.00%; p < 0.0001, ANOVA; Adjusted geometric mean (gMean) ratio = 102.33, 90% CI 2-sided [97.945 to 106.910], Standard Deviation 13.6 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax (Maximum Measured Concentration of Linagliptin Analyte in Plasma)
Description: This outcome measure presents maximum measured concentration of Linagliptin analyte in plasma.
  Time frame description: The time -1:00h was approximate; the procedure was to be performed and completed within 2h before drug administration. PKS including participants with available data for Cmax (maximum measured concentration of Linagliptin analyte in plasma).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | FDC (10 mg Empagliflozin and 5 mg Linagliptin) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets
Number analyzed (Participants) | 55 | 54
nmol/L | 9.33 (36.2) | 8.73 (37.1)
Statistical Analysis 1: Comparison: FDC (10 mg Empagliflozin and 5 mg Linagliptin) vs Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Bioequivalence acceptable range of 80.00% to 125.00%; p = 0.0027, ANOVA; Adjusted geometric mean (gMean) ratio = 107.51, 90% CI 2-sided [98.561 to 117.282], Standard Deviation 27.4 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of Empagliflozin in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: This outcome measure presents area under the concentration-time curve of Empagliflozin in plasma over the time interval from 0 extrapolated to infinity.
  Time frame description: The time -1:00h was approximate; the procedure was to be performed and completed within 2h before drug administration. PKS including participants with available data for AUC0-infinity (area under the concentration-time curve of Empagliflozin in plasma over the time interval from 0 extrapolated to infinity).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC (10 mg Empagliflozin and 5 mg Linagliptin) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets
Number analyzed (Participants) | 55 | 54
nmol*h/L | 2580 (18.0) | 2550 (19.8)
Statistical Analysis 1: Comparison: FDC (10 mg Empagliflozin and 5 mg Linagliptin) vs Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Adjusted geometric mean (gMean) ratio = 101.44, 90% CI 2-sided [99.574 to 103.336], Standard Deviation 5.7 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: This outcome measure presents area under the concentration-time curve of Linagliptin in plasma over the time interval from 0 extrapolated to infinity.
  Time frame description: The time -1:00h was approximate; the procedure was to be performed and completed within 2h before drug administration. PKS including participants with available data for (area under the concentration-time curve of Linagliptin in plasma over the time interval from 0 extrapolated to infinity).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC (10 mg Empagliflozin and 5 mg Linagliptin) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets
Number analyzed (Participants) | 55 | 54
nmol*h/L | 451 (25.9) | 462 (29.2)
Statistical Analysis 1: Comparison: FDC (10 mg Empagliflozin and 5 mg Linagliptin) vs Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Adjusted geometric mean (gMean) ratio = 98.15, 90% CI 2-sided [93.456 to 103.082], Standard Deviation 15.2 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 1 day after last drug administration, up to 77 days.
Arm/Group | FDC (10 mg Empagliflozin and 5 mg Linagliptin) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54
Other Adverse Events (participants affected / at risk) | 8/56 | 7/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDC (10 mg Empagliflozin and 5 mg Linagliptin) (N=56) | Empagliflozin (10 mg) + Linagliptin (5 mg) Single Tablets (N=54)
Headache (Nervous system disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No